CLINICAL TRIAL: NCT03423771
Title: An Exploratory Phase I/II Study on Safety, Pharmacokinetics and Efficacy of NPF-08 in Healthy Volunteers
Brief Title: Phase I/II Clinical Trial of NPF-08 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NPF-08-01/SE-01
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- NPF-08 Low dose （1-day treatment） (Experimental)
  Interventions: Drug: NPF-08
- NPF-08 Medium dose （2-day split dose） (Experimental)
  Interventions: Drug: NPF-08
- NPF-08 High dose （2-day split dose） (Experimental)
  Interventions: Drug: NPF-08
- NPF-08 Medium dose （1-day treatment） (Experimental)
  Interventions: Drug: NPF-08
- NPF-08 High dose （1-day treatment） (Experimental)
  Interventions: Drug: NPF-08
- NPF-08 Low～High dose （1-day treatment） (Experimental)
  Interventions: Drug: NPF-08
- NPF-08 Medium～High dose （2-day split dose） (Experimental)
  Interventions: Drug: NPF-08

INTERVENTIONS:
Drug: NPF-08 — Drug: NPF-08 Arms: NPF-08 oral sulfate solution

SUMMARY:
Japanese male healthy volunteers will receive NPF-08. The efficacy of NPF-08 will be assessed by intestinal cleaning degree. The safety of NPF-08 will be evaluated based on adverse events and adverse drug reactions observed from the date of administration to 7 days after administration.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy male volunteers (20 to 64 years old)
2. BMI（Body Mass Index）should be within a range of 17.6 and 26.4.
3. Subjects who agreed not to smoke or drink during hospital stay.
4. Subjects who do not excessively consume alcohol and those who do not excessively smoke
5. Subjects who are not judged as abnormal during the screening period in the physical examinations including 12-lead ECG, clinical symptoms, clinical examination, immunological examination (hepatitis B examination, hepatitis C examination, AIDS examination, syphilis examination).
6. Subjects who are not judged as abnormal during the before administration in blood electrolyte.
7. Subjects who have no clinical abnormalities and are judged to be eligible to the study by the investigator.

Exclusion Criteria:

1. Subjects who had previous significant gastrointestinal surgeries.
2. Subjects with a history of 12-lead ECG abnormality.
3. Subjects who have constipation（less than 2 bowel movement per week）
4. Subjects who have addictive of diarrhea
5. Subjects who have history of shock or hypersensitivity to sulfates (sodium sulfate, potassium sulfate, magnesium sulfate, etc.).
6. Subjects who have history of drug allergy.
7. Subjects who donated 200 mL or 400 mL of whole blood 4 weeks or 12 weeks respectively prior to the administration of investigational drug, or who donated blood component last 2 weeks.
8. Subjects who have participated in an investigational study within 4 months before signing the consent.
9. Subjects who is participating in the other investigational study
10. Subjects who received NPF-08 in the past
11. Subjects who are judged by the investigator as not adequate to participate the study.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Effective rate of overall intestinal cleaning effect (after washing of the observed region) by the Endoscopic Image Evaluation Committee (EIEC) | 1day

SECONDARY OUTCOMES:
Effective rate of overall intestinal cleaning effect (before washing of observed site) by EIEC | 1day
Cleaning effect by intestinal site (before/after washing of observed site) | 1day
Degree of bubbles by intestinal site | 1day
Time for completion of the bowel cleaning | 1day or 2day
Total dose of the investigational drug | 1day
Acceptability by subjects | up to 6hr
Coincidence rate of intestinal cleansing degree (before/after washing site of observation) between by EIEC members | 1day
Coincidence rate between the intestinal cleansing degrees evaluated by EIEC and the endoscope operators (before/after the observed site) | 1day

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Osaka, Japan